CLINICAL TRIAL: NCT02709018
Title: Enhancing Fear Extinction Via Angiotensin Type 1 Receptor Inhibition: A Randomized Controlled Trial in Posttraumatic Stress Disorder
Brief Title: A Controlled Trial of Losartan in Posttraumatic Stress Disorder
Acronym: LOSe-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Mclean Hospital (Other); Massachusetts General Hospital (Other); Henry M. Jackson Foundation, Walter Reed National Military Medical Center (Unknown); Foundation for Atlanta Veterans Education and Research, Inc. (Other); NYU Langone Health (Other); George Washington University (Other)
Responsible Party: Principal Investigator, Murray B. Stein, Professor of Psychiatry, Family Medicine and Public Health, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-15-2-0090
Record Dates: First submitted 2016-03-07; First posted 2016-03-15 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; losartan; angiotensin receptor blocker
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Experimental): Losartan flexibly dosed from 25-100 mg per day over 10 weeks
  Interventions: Drug: losartan
- Placebo (Placebo Comparator): Placebo flexibly dosed from 25-100 mg per day over 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: losartan — Angiotensin receptor blocker (ARB)
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to determine if losartan, an angiotensin receptor blocker (ARB), is safe and effective in the treatment of posttraumatic stress disorder (PTSD) symptoms. The study is also intended to determine if certain genetic markers are useful in predicting PTSD symptom reduction with losartan. Approximately 160 subjects with chronic PTSD ages 18-65 will participate in this study across five sites. Subjects will be assigned by chance to take either flexibly dosed losartan (up to a maximum dosage of 100 mg) or placebo (which resembles the study drug but has no active ingredients), once a day for 10 weeks. Furthermore, it is hypothesized that CC homozygotes for rs4311 SNP in the ACE gene will have a superior response to losartan on PTSD symptoms compared to T carriers.

DETAILED DESCRIPTION:
There are limited current treatments available for PTSD, and the only FDA-approved medications are SSRIs, which were empirically found to be somewhat helpful. Losartan provides a potentially important and exciting development in that it is readily available, safe, inexpensive (available as a generic drug), and has a neurobiological mechanism based on recent exciting discoveries, as outlined below. This proposal is designed to test, in a multisite RCT, this novel, mechanistically-determined, safe and well-tolerated, potentially powerful treatment for PTSD symptoms.

ELIGIBILITY:
[Below is a synopsis of relevant eligibility criteria. For details please refer to the protocol by contacting the Principal Investigator]

Inclusion Criteria

1. Subject must be a man or woman between 18 and 70 years of age, inclusive.
2. Subjects must have a primary DSM-5 diagnosis of Posttraumatic Stress Disorder.
3. Subjects must have a Clinical Administered PTSD Scale for PTSD (CAPS-5) ≥ 25 persistent at Screening for at least 3 months duration.
4. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
5. Subject must be willing and able to fill out self-administered questionnaires.
6. Subject must be able to be compliant with self-administration of medication.
7. Subject must be able to swallow the study medication whole with aid of water.
8. Subject must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria

1. Subjects who have current or imminent risk of suicide as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) at each study visit.
2. Subject with active psychosis.
3. Subject has a history of moderate or severe drug or alcohol use disorder according to DSM-5 criteria within 3 months before screening.
4. Subject has a history of allergy to losartan or other angiotensin receptor blockers (ARBs).
5. Subject has a medical illness likely to result in imminent hospitalization or for which treatments are contraindicated based on lab results, medical history and physical exam.
6. Subject has serious cognitive impairment felt likely to interfere with the ability to participate meaningfully in the study. Participants with mild to moderate traumatic brain injury (TBI) will not be excluded from the study. Only those who evidence significant cognitive impairment at Screening (as evidenced by confusion, inability to track discussion or answer questions, or other clear and significant indicators of cognitive impairment) will be excluded.
7. Concurrent ACE Inhibitors or Angiotensin Receptor Blockers or Prazosin; patients on other antihypertensives may be enrolled if, after consultation with their prescribing physician, it is determined that the addition of losartan would not be contraindicated.
8. Concurrent antidepressants or antipsychotics. Subjects, who have elected, in consultation with their health care provider, to discontinue any antidepressants or antipsychotics, must be off the medications for a minimum of 2 weeks prior to study randomization. Stable bedtime doses of sleep agents (e.g., trazodone ≤ 200mg; eszopiclone; zolpidem; lorazepam) will be allowed as long as the dose has been stable for at least 2 weeks prior to study randomization. Benzodiazepines taken for other than sleep are not permitted.
9. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant.
10. Subject is unable to comply with the study-specific requirements
11. Subjects with abnormal liver, renal or EKG findings as determined by physician.
12. Subject exhibits clinically-significant hypertension as determined by medical evaluation and/or BP > 190/100.
13. Systolic Blood Pressure (SBP) < 90mmHg.
14. Liver function Tests (LFT's) > 2 times the upper limit of normal.
15. Patients with Chronic Kidney Disease 4, as determined by history, baseline labs (including eGFR < 45ml/minute) and evaluation by a physician will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-07-16 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD, MPH, Principal Investigator — University of California, San Diego; Kerry J Ressler, MD, PhD, Study Chair — McLean Hospital and Harvard Medical School
Locations (6):
- United States (6):
  - University of California, San Diego, La Jolla, California
  - George Washington University, Washington D.C., District of Columbia
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khoury NM, Marvar PJ, Gillespie CF, Wingo A, Schwartz A, Bradley B, Kramer M, Ressler KJ. The renin-angiotensin pathway in posttraumatic stress disorder: angiotensin-converting enzyme inhibitors and angiotensin receptor blockers are associated with fewer traumatic stress symptoms. J Clin Psychiatry. 2012 Jun;73(6):849-55. doi: 10.4088/JCP.11m07316. Epub 2012 May 1. PMID 22687631
- [Background] Krause EG, de Kloet AD, Scott KA, Flak JN, Jones K, Smeltzer MD, Ulrich-Lai YM, Woods SC, Wilson SP, Reagan LP, Herman JP, Sakai RR. Blood-borne angiotensin II acts in the brain to influence behavioral and endocrine responses to psychogenic stress. J Neurosci. 2011 Oct 19;31(42):15009-15. doi: 10.1523/JNEUROSCI.0892-11.2011. PMID 22016534
- [Background] Llano Lopez LH, Caif F, Garcia S, Fraile M, Landa AI, Baiardi G, Lafuente JV, Braszko JJ, Bregonzio C, Gargiulo PA. Anxiolytic-like effect of losartan injected into amygdala of the acutely stressed rats. Pharmacol Rep. 2012;64(1):54-63. doi: 10.1016/s1734-1140(12)70730-2. PMID 22580520
- [Background] Saavedra JM, Sanchez-Lemus E, Benicky J. Blockade of brain angiotensin II AT1 receptors ameliorates stress, anxiety, brain inflammation and ischemia: Therapeutic implications. Psychoneuroendocrinology. 2011 Jan;36(1):1-18. doi: 10.1016/j.psyneuen.2010.10.001. Epub 2010 Oct 29. PMID 21035950
- [Background] Nylocks KM, Michopoulos V, Rothbaum AO, Almli L, Gillespie CF, Wingo A, Schwartz AC, Habib L, Gamwell KL, Marvar PJ, Bradley B, Ressler KJ. An angiotensin-converting enzyme (ACE) polymorphism may mitigate the effects of angiotensin-pathway medications on posttraumatic stress symptoms. Am J Med Genet B Neuropsychiatr Genet. 2015 Jun;168B(4):307-15. doi: 10.1002/ajmg.b.32313. Epub 2015 Apr 29. PMID 25921615
- [Background] Hurt RC, Garrett JC, Keifer OP Jr, Linares A, Couling L, Speth RC, Ressler KJ, Marvar PJ. Angiotensin type 1a receptors on corticotropin-releasing factor neurons contribute to the expression of conditioned fear. Genes Brain Behav. 2015 Sep;14(7):526-33. doi: 10.1111/gbb.12235. Epub 2015 Aug 25. PMID 26257395
- [Background] Marvar PJ, Goodman J, Fuchs S, Choi DC, Banerjee S, Ressler KJ. Angiotensin type 1 receptor inhibition enhances the extinction of fear memory. Biol Psychiatry. 2014 Jun 1;75(11):864-72. doi: 10.1016/j.biopsych.2013.08.024. Epub 2013 Oct 4. PMID 24094510
- [Derived] Stein MB, Jain S, Simon NM, West JC, Marvar PJ, Bui E, He F, Benedek DM, Cassano P, Griffith JL, Howlett J, Malgaroli M, Melaragno A, Seligowski AV, Shu IW, Song S, Szuhany K, Taylor CT, Ressler KJ; LOSe-PTSD Investigators. Randomized, Placebo-Controlled Trial of the Angiotensin Receptor Antagonist Losartan for Posttraumatic Stress Disorder. Biol Psychiatry. 2021 Oct 1;90(7):473-481. doi: 10.1016/j.biopsych.2021.05.012. Epub 2021 May 21. PMID 34275593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 75 | 74
Completed | 59 | 58
Not Completed | 16 | 16

BASELINE CHARACTERISTICS:
Population: The primary outcome (CAPS-5) was analyzed using an MMRM (mixed model repeated measures) approach based on a modified intent-to-treat (mITT) population, defined as randomized subjects who initiated treatment and had both a baseline and at least one post-baseline outcome score during the blinded phase of the study (Week 10). Participants from the mITT population who were included in the MMRM model also required both a baseline and at least one post-baseline CAPS-5 score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (12.3) | 35.5 (12.6) | 36.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 54 | 97
  Male | 32 | 20 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 14 | 22
  White | 50 | 44 | 94
  More than one race | 6 | 11 | 17
  Unknown or Not Reported | 1 | 2 | 3
CAPS-5 Total [Mean (Standard Deviation); unit: units on a scale] — The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) score as administered here reflects the sum of the 20 DSM-5 PTSD items, each scored 0-4. Range of the scale is 0-80. Higher scores indicate greater severity.
  units on a scale | 33.5 (10.3) | 34.2 (10.0) | 33.8 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome for This Study is Mean Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Over the Treatment Period of 10 Weeks Between the Losartan Arm and the Placebo Arm.
Description: Clinician-Administered PTSD Scale for DSM-5 also known as CAPS-5 is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to, make current (past month) diagnosis of PTSD, make a lifetime diagnosis of PTSD and assess PTSD symptoms over the past week.
  The CAPS-5 as used here has 20 items, each scored 0-4, to yield a score with a possible range of 0-80. Higher scores mean worse outcome.
Time Frame: 10 weeks
Population: Modified Intent to Treat (mITT) Population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 58 | 58
score on a scale | -15.96 [-18.86 to -13.06] | -16.89 [-19.81 to -13.97]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority; p = 0.66, Mixed Models Analysis

2. Secondary Outcome: Change in CAPS-5 Associated With CC Homozygosity for rs4311 SNP in the Angiotensin Converting Enzyme Gene (ACE) Compared to T Carriers, Among Subjects Randomized to Losartan.
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) as used here has 20 items, each scored 0-4, to yield a score with a possible range of 0-80. Higher scores mean worse outcome.
Time Frame: 10 weeks
Population: Subjects on Losartan Arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CC Homozygotes on Losartan: CC Homozygotes on Losartan
- T Carriers on Losartan: T Carriers on Losartan
Arm/Group | CC Homozygotes on Losartan | T Carriers on Losartan
Number analyzed (Participants) | 11 | 40
score on a scale | 16.7 (10.1) | 15.8 (13.1)
Statistical Analysis 1: Comparison: CC Homozygotes on Losartan vs T Carriers on Losartan; Test type: Superiority; p = 0.57, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 10 Weeks (Study Duration)
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 2/75 | 1/74
Other Adverse Events (participants affected / at risk) | 20/75 | 18/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=75) | Placebo (N=74)
Neurosyphilis (Nervous system disorders) | 0 (0) | 1 (1) — Neurosyphilis not reported at baseline but reported during study
Cataplexy (Nervous system disorders) | 1 (1) | 0 (0)
Gallbladder Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=75) | Placebo (N=74)
Lightheadedness (Nervous system disorders) | 8 (13) | 7 (9)
Insomnia (Nervous system disorders) | 4 (4) | 5 (5)
headache (Nervous system disorders) | 16 (24) | 14 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT02709018/Prot_SAP_000.pdf